CLINICAL TRIAL: NCT02920320
Title: iCompassion: Internet-based Self-help for More Self-compassion
Acronym: iCompassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TK001
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Self-criticism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based self-help (Experimental): Internet-based self-help on the basis of the program "Mindfulness-Based Compassionate Living" (van den Brink & Koster, 2015). The self-help program consists of seven text-based sessions, various exercises (z.B. breathing meditations, diaries,) and tasks. Participants have the possibility for guidance to the program on request.
  Interventions: Other: Internet-based self-help program
- Waiting control group (No Intervention)

INTERVENTIONS:
Other: Internet-based self-help program
  Arms: Internet-based self-help

SUMMARY:
In this study, people who suffer from strong self-critical tendencies will be randomized to two study conditions. The first group receives an account to an internet-based self-help intervention. The second group is a waiting control group. In both conditions additional care or treatment is allowed. The aim of the study is to investigate the effectiveness of an internet-based self-help intervention on depressive, anxiety and stress symptoms compared to a waiting list. Assessments are at baseline, 8-week and 6-months post-randomization. After 8 weeks, participants in the waiting control group get also access to the intervention and fill out questionnaires after 8 weeks again.

ELIGIBILITY:
Inclusion Criteria:

* Increased levels of self-criticism
* 18 years or older
* Internet account
* Sufficient German language skills
* Written informed consent

Exclusion Criteria:

* Substance dependence, psychotic disorder, bipolar disorder
* Acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Depression anxiety stress scale (DASS) | 8-week

SECONDARY OUTCOMES:
Self-Compassion Scale | Baseline, 8-week, 6-month
Mini International Neuropsychiatric Interview | Baseline, 8-week
Forms of Self-Criticism and Self-Reassurance Scale | Baseline, 8-week, 6-month
Comprehensive Inventory of Mindfulness Experiences | Baseline, 8-week, 6-month
Positive and Negative Affective Schedule | Baseline, 8-week, 6-month
Fear of Self-Compassion Scale | Baseline, 8-week, 6-month
Satisfaction with Life Scale | Baseline, 8-week, 6-month
Questionnaire for the Assessment of Adaptive and Maladaptive Shame | Baseline, 8-week, 6-month
Rosenberg Self-Esteem Scale | Baseline, 8-week, 6-month follow-up
Client Satisfaction Questionnaire | 8-week
Depression anxiety stress scale (DASS) | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Krieger, PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided